CLINICAL TRIAL: NCT06517693
Title: Open-Label, Phase I Study of the Safety and Pharmacokinetics of PGT121.414.LS Alone and in Combination With VRC07-523LS in Infants Exposed to HIV-1
Brief Title: Safety and Pharmacokinetics Study of PGT121.414.LS Alone and in Combination With VRC07-523LS in Infants Exposed to HIV-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute of Allergy and Infectious Diseases Vaccine Research Center (NIAID VRC) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IMPAACT 2037; 38962 (Other: DAIDS Study ID)
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HIV-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Stratum Formula Fed (FF) (Experimental): Single subcutaneous (SC) dose of PGT121.414.LS at birth, based on weight.
  Interventions: Drug: PGT121.414.LS
- Cohort 1 Stratum Breastfed (BF) (Experimental): Initial SC dose of PGT121.414.LS at birth, based on weight. Second SC dose of 100 mg PGT121.414.LS at Week 12, if still breastfeeding. Dosing at Week 12 is not based on weight.
  Interventions: Drug: PGT121.414.LS
- Cohort 2 Stratum FF (Experimental): Single SC doses of PGT121.414.LS and VRC07-523LS at birth, based on weight.
  Interventions: Drug: PGT121.414.LS; Drug: VRC07-523LS
- Cohort 2 Stratum BF (Experimental): Initial SC doses of PGT121.414.LS and VRC07-523LS at birth, based on weight. Second SC doses of 100 mg of PGT121.414.LS and 100 mg VRC07-523LS at Week 12, if still breastfeeding. Dosing at Week 12 is not based on weight.
  Interventions: Drug: PGT121.414.LS; Drug: VRC07-523LS

INTERVENTIONS:
Drug: PGT121.414.LS — Administered SC in the thigh
Drug: VRC07-523LS — Administered SC in the thigh
  Arms: Cohort 2 Stratum BF; Cohort 2 Stratum FF

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics (PK) of the potent, broadly neutralizing anti-HIV monoclonal antibodies (mAb) PGT121.414.LS alone and in combination with VRC07-523LS soon after birth in infants exposed to HIV-1.

DETAILED DESCRIPTION:
This is an open-label, phase I study of the potent, broadly neutralizing anti-HIV monoclonal antibodies (mAb) PGT121.414.LS alone and in combination with VRC07-523LS administered soon after birth in infants exposed to HIV-1. The study is designed to assess the safety and pharmacokinetics (PK) profile of one and two subcutaneous (SC) doses of PGT121.414.LS alone or in combination with VRC07-523LS through Week 12 and Week 24, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Birthing parent is of legal age or circumstance to provide independent informed consent and is willing and able to provide written informed consent for themselves and permission for their infant's participation in this study.
* Birthing parent has confirmed HIV-1 infection based on positive test results from two samples collected from two separate blood collection tubes.
* Infant was singleton or twin.
* Infant's gestational age at birth was at least 36 weeks.
* At birth, infant's weight was at least 2 kg.
* At entry, infant is less than 72 hours of age and is anticipated to receive study product within 72 hours after birth.
* At screening, infant has the following laboratory test results:

  * Hemoglobin, normal or grade 1 (≥13 g/dL or ≥8.05 mmol/L)
  * Platelets, normal or grade 1 (≥100,000 cells/mm3 or ≥100.000 x10^9 cells/L)
  * Absolute neutrophil count (ANC), normal or grade 1

    1. ≤24 hours old (≥4,000 cells/mm3 or ≥4.000 x10^9 cells/L)
    2. >24 hours old (≥1,250 cells/mm3 or ≥1.250 x10^9 cells/L)
  * Alanine transaminase (ALT), normal (<1.25 x ULN)
* At entry, infant is generally healthy as determined by the site investigator based on review of all available medical history information and physical examination findings.
* Cohorts 1 and 2, Strata BF only: At entry, infant is breastfeeding or the birthing parent has indicated an intention to initiate breastfeeding.
* Cohorts 1 and 2, Strata FF, only: At entry, infant is not breastfeeding and the birthing parent has indicated no intention to breastfeed.
* At entry, infant is at increased risk of HIV acquisition.

Cohorts 1 and 2, Strata FF only:

* Birthing parent had acute HIV during this pregnancy; or
* Birthing parent with detectable viral replication (plasma HIV RNA results at least 50 copies/mL) during pregnancy who did not have confirmed viral suppression, defined as at least two consecutive plasma HIV RNA results less than 50 copies/mL from specimens obtained at least four weeks apart with the latest result within four weeks prior to delivery; or
* Birthing parent not receiving appropriate ART for at least two weeks, with any part of the two-week period occurring within four weeks prior to delivery, based on birthing parent's report or available medical records.

Cohorts 1 and 2, BF only:

* Per birthing parent's report, intends to breastfeed

Exclusion Criteria:

* Birthing parent has received any investigational product during this pregnancy.
* Infant has received any active or passive HIV immunotherapy or any investigational product.
* At entry, infant with a documented positive HIV Nucleic Acid Test (NAT) result.
* Birthing parent or infant has any condition that, in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants with at least one Grade 3 or higher Adverse Event (AE) (one dose) | Day 0 through Week 12
Proportion of infants with at least one Grade 3 or higher AE assessed as related to study product (one dose) | Day 0 through Week 12
Proportion of infants with at least one Grade 3 or higher AE (two doses) | Day 0 through Week 24
Proportion of infants with at least one Grade 3 or higher AE assessed as related to study product (two doses) | Day 0 through Week 24
PGT121.414.LS maximum concentration (Cmax) (single/first dose) | Day 0 through Week 48
PGT121.414.LS time of maximum concentration (Tmax) (single/first dose) | Day 0 through Week 48
PGT121.414.LS area under the curve (AUC(0-12WK)) (single/first dose) | Day 0 through Week 12
PGT121.414.LS concentration at the end of the first dose interval (C(12WK)) (single/first dose) | Week 12
PGT121.414.LS concentration at the end of the second dose interval (C(24WK)) (two doses) | Week 24
VRC07-523LS maximum concentration (Cmax) (single/first dose) | Day 0 through Week 48
VRC07-523LS time of maximum concentration (Tmax) (single/first dose) | Day 0 through Week 48
VRC07-523LS area under the curve (AUC(0-12WK)) | Day 0 through Week 12
VRC07-523LS concentration at the end of the first dose interval (C(12WK)) single/first dose) | Week 12
VRC07-523LS concentration at the end of the second dose interval (C(24WK)) (two doses) | Week 24

SECONDARY OUTCOMES:
Proportion of infants with at least one Grade 3 or higher AE | Day 0 through Week 96
Proportion of infants with at least one Grade 3 or higher AE assessed as related to study product | Day 0 through Week 96
Proportion of infants with at least one Grade 2 or higher AE (one dose) | Day 0 through Week 12
Proportion of infants with at least one Grade 2 or higher AE assessed as related to study product (one dose) | Day 0 through Week 12
Proportion of infants with at least one Grade 2 or higher AE (two doses) | Day 0 through Week 24
Proportion of infants with at least one Grade 2 or higher AE assessed as related to study product (two doses) | Day 0 through Week 24
Proportion of infants with any AEs that lead to study product discontinuation | Day 0 through Week 12
PGT121.414.LS AUC(0-48WK) after single dose administration | Week 48
PGT121.414.LS concentration after single dose administration | Week 48
PGT121.414.LS concentration after two dose administration | Week 60
PGT121.414.LS apparent clearance (CL/F) | Day 0 through Week 60
PGT121.414.LS half-life (T1/2) following single dose administration | Day 0 through Week 48
PGT121.414.LS half-life (T1/2) following two dose administration | Day 0 through Week 60
VRC07-523LS AUC(0-48WK) after single dose administration | Week 48
VRC07-523LS concentration after single dose administration | Week 48
VRC07-523LS concentration after two dose administration | Week 60
VRC07-523LS apparent clearance (CL/F) | Day 0 through Week 60
VRC07-523LS half-life (T1/2) following single dose administration | Day 0 through Week 48
VRC07-523LS half-life (T1/2) following tow dose administration | Day 0 through Week 60
Proportion of infants with PGT121.414.LS concentrations > 20 and > 50 mcg/mL following single/first dose administration | Week 12
Proportion of infants with PGT121.414.LS concentrations > 20 and > 50 mcg/mL following two dose administration | Week 24
Proportion of infants with VRC07-523LS concentrations > 10 and > 20 mcg/mL following single/first dose administration | Week 12
Proportion of infants with PGT121.414.LS concentrations > 10 and > 20 mcg/mL following two dose administration | Week 24
Proportion of infants with anti-PGT121.414.LS antibodies detected | Week 24
Proportion of infants with anti-VRC07-523LS antibodies detected | Week 24
Proportion of infants with anti-PGT121.414.LS antibodies detected | Week 48
Proportion of infants with anti-VRC07-523LS antibodies detected | Week 48
Proportion of infants with confirmed HIV infection following receipt of study product | Day 0 through Week 96
Frequency of study product injection site local reactions for one and two SC doses of PGT121.414.LS alone or in combination with VRC07-523LS | Day 0 through Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Coleen Cunningham, Study Chair — University of California, Irvine
Locations (16):
- United States (11):
  - Site 5112, David Geffen School of Medicine at UCLA, Los Angeles, California
  - Site 5052, University of Colorado Denver, Aurora, Colorado
  - Site 5051, University of Florida Jacksonville, Jacksonville, Florida
  - Site 5127, Pediatric Perinatal HIV, Miami, Florida
  - Site 5030, Emory University School of Medicine, Atlanta, Georgia
  - Site 5083, Rush University Cook County Hospital Chicago, Chicago, Illinois
  - Site 5092, Johns Hopkins University Baltimore, Baltimore, Maryland
  - Site 5114, Bronx-Lebanon Hospital Center, The Bronx, New York
  - Site 5013, Jacobi Medical Center Bronx, The Bronx, New York
  - Site 6501, St. Jude Children's Research Hospital, Memphis, Tennessee
  - Site 5128, Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
- Brazil (2):
  - Site 5072, Hospital Federal dos Servidores do Estado, Rio de Janeiro
  - Site 5097, Hospital Geral De Nova Iguacu Brazil, Rio de Janeiro
- Site 5121, Kenya Medical Research Institute/Walter Reed Project Clinical Research Center, Kericho, Kericho, Kenya
- Site 5129, IMPAACT/Gamma Project/UPR Pediatric HIV/AIDS Research, San Juan, Puerto Rico
- Site 8950, FAMCRU, Cape Town, Parrow Valley, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: With whom?
  * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
  * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
  * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https:// www.impaactnetwork.org/ resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: https://www.impaactnetwork.org/studies/impaact2037